CLINICAL TRIAL: NCT04622722
Title: Efficacy and Safety of Diabetes-specific Formula in Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Collaborators: Ramathibodi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 18.01.TH.CLI
Record Dates: First submitted 2018-12-06; First posted 2020-11-10 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-10

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes-specific formula
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: This is an open-label, randomized cross-over study.
  The study date will be 1 day for group A and 1 day for group B, separated by 7-day wash out period.
  The tolerability of DSF, assessed by questionnaire, will be collected while the subjects consume DSFs daily 7 days before the study date (only group A). The questionnaire will ask about gastrointestinal symptom including abdominal distention, nausea, vomiting, and stool frequency.
  Group A participants will be asked to drink 360 ml of Nutren Diabetes which provides 360 kcal.
  Group B participants will be asked to consume isocaloric diet (360 kcal)comprising one carton of soy milk (250 ml) and bologna and mayonnaise sandwiches (two slices of bread).
  Plasma glucose and insulin will be collected at baseline (minute 0) and 30, 60, 120 minute postprandially. The participants will be asked to complete the questionnaire (Visual analog scale) to assess hunger and satiety at minute 0, 30, 60 and 120 minute.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Group A: Drinking Nutren Diabetes provides energy at 360 kcal per 360 ml
  Interventions: Other: Nutren Diabetes; Other: Isocaloric
- Group B (Placebo Comparator): Group B: Having Isocaloric diet provide 360 kcal.
  Interventions: Other: Nutren Diabetes; Other: Isocaloric

INTERVENTIONS:
Other: Nutren Diabetes — Nutren Diabetes provides energy at 360 kcal per 360 ml
Other: Isocaloric — Isocaloric diet One carton of soy milk (250 ml) and bologna sandwiches (two slices of bread) with mayonnaise

SUMMARY:
Hypothesis: the diabetes-specific formula Nutren diabetes provides better postprandial glucose control in patients with type 2 diabetes when compared to the isocaloric diet.

DETAILED DESCRIPTION:
This study is an open label, randomized controlled cross-over study

Research objectives:

1. To study the efficacy of diabetes-specific formula (Nutren Diabetes) in comparison with an isocaloric diet in the aspect of postprandial blood glucose and insulin response (baseline, 30, 60 and 120 minute).
2. To study the safety and tolerance of a diabetes-specific formula compared with an isocaloric diet in patients with type 2 diabetes mellitus

Statistical analysis method

1. Descriptive statistics: categorical data will be summarized as number and percentage, continuous data with normal distribution will be presented as means and standard deviations, and continuous data with non-normal distribution will be summarized as median, minimum and maximum.
2. Inferential statistics: Repeated Measure ANOVA from analyzing the difference of means from measuring fasting glucose and insulin more than two times.
3. Inferential statistics: Paired T-Test or Wilcoxon Matched pairs Signed Rank Test derived by analyzing the comparison between the means of two dependent groups.
4. Report of the difference between two categories by the difference of means with 95% Confidence Interval
5. Number of participant (subjects) and criteria for participation 30 participants by calculation formula of Frison and Pocock (1992) with STATA program.

ELIGIBILITY:
Inclusion Criteria:

* DM type 2, HbA1C < 9% FPG < 180 mg/dl
* Aged between 18- 70 years.
* Participants must have stable body weight (+/- not over 5%) for the past six months.
* Participants must control their diabetes by diet control or taking diabetes medicine without medicine dose adjustment during the period of the research.
* Participants are willing to participate in the research and sign written consent form.

Exclusion Criteria:

* Participants receive insulin hormone and GPL-1 agonist injection.
* GFR < 30 ml/min/1.73 m2
* Participants have decompensated liver cirrhosis or alcoholism or drug abuse record.
* Participants have record of allergy to any ingredients in diabetes-specific formula,soybean milk or bologna and mayonnaise sandwich.
* Participants decline to participate

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-08-22 (Actual); Primary Completion 2020-05-16 (Actual); Study Completion 2020-05-16 (Actual)

PRIMARY OUTCOMES:
2-hour postprandial glucose | Change form baseline blood glucose level at 30,60, and 120 min.
  The primary outcome will be the difference of 2-hour postprandial glucose between group A and group B

SECONDARY OUTCOMES:
Area under the curve of postprandial plasma glucose (AUC glucose 0-120 min) | Time Frame: Postprandial blood glucose response at 0, 30, 60,120 min
  The secondary outcome will be the difference of AUC glucose 0-120 min between group A and group B.
  Blood samples will be collected to assess plasma glucose at baseline and 30, 60, 120-minute postprandial. We will calculate the area under the curve of plasma glucose of patients in each arm at baseline and, 30, 60, 120 minute postprandial (AUC glucose 0-120 min) .
  Blood samples will be collected to assess plasma insulin at baseline and 30, 60, 120-minute postprandial. We will calculate the area under the curve of plasma insulin of patients in each arm at baseline and, 30, 60, 120 minute postprandial (AUC insulin 0-120 min) .
Area under the curve of postprandial plasma insulin (AUC insulin 0-120 min) | Postprandial plasma insulin response at 0, 30, 60,120 min
  The secondary outcome will be the difference of AUC insulin 0-120 min between group A and group B.
Gastrointestinal tolerance | 7 days prior to the treatment phase.
  Gastrointestinal tolerance including abdominal distention, nausea, vomiting, and stool frequency will be assessed by questionnaire. We will collect the symptom of GI tolerance everyday during the period that the patient consumes Nutren diabetes and isocaloric diet (7 days before the study date; only participants in group A )

CONTACTS AND LOCATIONS:
Overall Officials: Daruneewan Warodomwichit, Principal Investigator — Division of Nutrition & Biochemical Medicine, Department of Medicine
Locations (1):
- Division of Nutrition & Biochemical Medicine, Department of Medicine, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gulati S, Misra A, Nanda K, Pandey RM, Garg V, Ganguly S, Cheung L. Efficacy and tolerance of a diabetes specific formula in patients with type 2 diabetes mellitus: An open label, randomized, crossover study. Diabetes Metab Syndr. 2015 Oct-Dec;9(4):252-7. doi: 10.1016/j.dsx.2014.10.001. Epub 2014 Nov 1. PMID 25458669